CLINICAL TRIAL: NCT06590441
Title: A Multisite Investigation of the Wearing Compliance of Spectacles for Myopia Control
Brief Title: Investigation of Wearing Compliance of Spectacles for Myopia Control
Status: Completed | Type: Observational
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Other Study IDs: EX-MKTG-160
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Myopia control spectacle wearers: Established (use of ≥3 months) juvenile myopia control spectacle wearers
  Interventions: Device: Myopia control spectacles

INTERVENTIONS:
Device: Myopia control spectacles — Myopia control spectacles fitted with temperature sensors

SUMMARY:
The goal of this observational study was to compare the wearing patterns of spectacles prescribed for myopia control in juvenile wearers.

DETAILED DESCRIPTION:
This unmasked, multi-center, observational study evaluated the wearing patterns of established (use of ≥3 months) juvenile spectacles wearers. It aimed to compare the wearing patterns of spectacles for myopia control between males and females. Wearing pattern were measured via the use of temperature sensors fitted to the sides of the participant's spectacles. Data from the final week of the 1-month study was used for analysis to minimize 'unusual' wear patterns which may have occurred early in the study.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged between six and 15 years old.
2. Their parent or guardian understands the rights of the subject and are willing to sign a statement of informed consent.
3. They understand the study at a level appropriate for their age and are willing to sign a statement of assent.
4. They and their parents or guardians are willing and able to follow the protocol.
5. They currently use spectacle lenses for myopia control and have done so for at least three months.
6. They agree not to participate in other clinical research for the duration of this study.

Exclusion Criteria:

1. They have an unusual ophthalmic history, which in the opinion of the site investigator or Principal Investigator might impact on the successful conduct of the study.
2. They are amblyopic.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Juvenile participants recruited directly from the patient bases of several UK optometry practices who currently wear spectacles prescribed for myopia
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, Principal Investigator — Eurolens Research
Locations (4):
- United Kingdom (4):
  - Eye2C Ltd, Sale, Cheshire
  - Susan Hilton Ltd, Darwen, England
  - Columbo Ltd, Oakwood, Leeds
  - David Gould Opticians Limited, Haslingden, Rossendale

RESULTS

PARTICIPANT FLOW:
Groups:
- Myopia Control Spectacles: All participants wore their habitual myopia control spectacles
Period: Overall Study
Arm/Group | Myopia Control Spectacles
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Myopia Control Spectacles: All participants of the clinical study
Arm/Group | Myopia Control Spectacles
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Wearing Pattern of Myopia Control Spectacles
Description: Overall wearing patterns were evaluated via the use of temperature sensors fitted to the frame of the spectacles. The temperature readings from the final week of the one month study were used to determine when spectacles were worn or removed. Scores were calculated as the average times over a 24 hour period (W24) where a higher score indicated that the spectacles were worn for a longer period of time per day.
Time Frame: Measured continuously over 1 week of wear
Population: Data for one participant was not available due to a failure of the sensors
Measure: Mean (Standard Deviation); unit: Hours in a day
Groups:
- Myopia Control Spectacles: Participants that wore habitual myopia control spectacles with fully working sensors
Arm/Group | Myopia Control Spectacles
Number analyzed (Participants) | 52
Hours in a day | 12.8 (4.1)

2. Primary Outcome: Effect of Sex on Overall Wearing Pattern
Description: The effect of sex on the overall wearing pattern was evaluated via the use of temperature sensors fitted to the frame of the spectacles. The temperature readings from the final week of the one month study were used to determine when spectacles were worn or removed. Scores were calculated as the average times over a 24 hour period (W24) and a 'waking day' period of 07:00 to 21:00 (W14), where a higher score indicated that the spectacles were worn for a longer period of time per day.
Time Frame: Measured continuously over 1 week of wear
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours in a day
Groups:
- Female Participants: Female participants that wore habitual myopia control spectacles with fully working sensors
- Male Participants: Male participants that wore habitual myopia control spectacles with fully working sensors
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 29 | 23
Hours in a day
  W14 | 12 [11.0 to 13.0] | 10.4 [9.2 to 11.5]
  W24 | 13.9 [12.6 to 15.1] | 11.5 [10.1 to 12.9]

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately one month.
Arm/Group | Myopia Control Spectacles
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT06590441/Prot_SAP_000.pdf